CLINICAL TRIAL: NCT00628680
Title: Pivotal/Phase III Multicentered, Two-Arm, Randomized Study Comparing the Effects of AAT-023 Solution (Zuragen), and Heparin on the Incidence of Catheter Related Blood Stream Infections in Tunneled Chronic Central Venous Catheters for Dialysis
Brief Title: A Multi-Centered, Two-Arm, Randomized Study Comparing the Effects of AAT-023 (Zuragen) Solution, and Heparin on the Incidence of Catheter Related Blood Stream Infections in Tunneled Chronic Central Venous Catheters for Dialysis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ash Access Technology (Industry)
Responsible Party: Roland Winger, VP of Clinical and Product Development, Ash Access Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AATML2003-A
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: End Stage Renal Disease
Keywords: Renal Disease; Kidney Failure; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Renal Insufficiency | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AAT-023 (Zuragen Arm) (Experimental): Active experimental consisting of AAT-023 (Zuragen)solution
  Interventions: Device: AAT-023 solution (Zuragen)
- Heparin (Active Comparator): 5000 units diluted with normal saline to the exact catheter lumen volume
  Interventions: Drug: Heparin

INTERVENTIONS:
Device: AAT-023 solution (Zuragen) — Amount equal to the catheter lumen plus 0.3mL. Three times per week (after each Hemodialysis) for 26 weeks
  Arms: AAT-023 (Zuragen Arm)
Drug: Heparin — Hepaarin 5000 units diluted with normal saline to the exact catheter lumen volume.
  Arms: Heparin

SUMMARY:
The purpose of this study is to determine if AAT-023 (Zuragen) solution is superior to Heparin in preventing Catheter Related Blood Stream Infections for End Stage Renal Disease patients.

DETAILED DESCRIPTION:
The purpose of this study is to show that AAT-023 (Zuragen) Solution is superior to Heparin in preventing Catheter Related Blood Stream Infections (CRBSI) when used as a catheter lock solution in Central Venous Catheter's for Dialysis between hemodialysis treatments (3x per week), where CRBSI's are defined as concordant bacteria found in both the catheter and peripheral blood or the exit site and peripheral blood in subjects demonstrating a temperature greater than 38 degrees celcius.

ELIGIBILITY:
Inclusion Criteria:

1. End Stage Renal Disease 18 yrs or older.
2. CVCD with average dialysis flow rate over 300 mL/min for three most recent visits.
3. Expectation by Investigator that CVCD may be needed for up to 26 weeks.
4. Dialysis catheter is of three types a) single body with single entry and exit, b) single body with split ends, c) twin catheter with one catheter for removal of blood and another for return.
5. Kt/V >1.1 or equivalent URR
6. Negative serum pregnancy unless surgically sterile or post menopausal for >1yr.
7. Negative blood culture result from pre-enrollment blood sample draw.
8. Ability of patient to sign and understand the informed consent.
9. Most recent lab results don't indicate hypocalcemia (<7mg/dL) or thrombocytopenia (<20,000)
10. Avg. systolic blood pressure >90 mmHg as measured during the most recent three dialysis treatments.
11. Lack of signs of current blood stream infection at the beginning of the prior three dialysis treatments.

Exclusion Criteria:

1. A known Heparin allergy or a history of type 2 (antibody mediated) Heparin-induced thrombocytopenia.
2. Active bleeding from any site or a documented positive stool hemocult test within 28 days of enrollment in study.
3. Bloodstream infection,exit site infection or any infection requiring antibiotic use within 14 days of enrollment for any antibiotic listed in section 4.2.3 or within 30 days of enrollment for Vancomycin or any other antibiotic not listed in section 4.2.3 of the protocol
4. Inability to comply with the conditions of, or complete the protocol in the opinion of the Investigator.
5. Pregnant or breast feeding.
6. Documented allergy to sodium citrate, methylene blue, methyl/paraben and/or propyl paraben.
7. Documented chronic intrinsic coagulopathy evidenced by persistently and significantly elevated Prothrombin (INR>3), Partial Thromboplastin Time (PTT>60 seconds), or thrombocytopenia (platlet count <20,000/mm).
8. Malignancy requiring chemotherapy or radiation treatment within 180 days of enrollment.
9. Documented requirement for >5,000 units of Heparin per catheter lumen to maintain catheter patency (with decrease in blood flow demonstrated at 5,000 units per lumen Heparin catheter lock) with current catheter.
10. Contraindications to citrate or taking drugs that may interact with citrate.
11. Documented history of glucose-6-phosphate dehydrogenase deficiency (G6PD or Drug-induced methemoglobinemia).
12. Participation in another research study.
13. Co-morbidities, such as HIV, active hepatitis or recent transplants, that in the opinion of the Investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results and would make the subject inappropriate for entry into this study.
14. Unknown priming volume of catheter lumens.
15. Redness of over 1 cm diameter or pus around the catheter exit site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To show that AAT-023 (Zuragen) solution is superior to Heparin in preventing CRBSI when used as a catheter lock solution in CVCD's between hemodialysis treatments. | 6 months

SECONDARY OUTCOMES:
To show that AAT-023 (Zuragen) solution is non-inferior to Heparin in terms of patency failure. | 6 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Bakersfield Dialysis Center, Bakersfield, California
  - Renal Medical Associates, Lynwood, California
  - Nephrology & Hypertension Associates, PC, Middlebury, Connecticut
  - Brandon nephrology, Brandon, Florida
  - Gulf Breeze Dialysis Center, Dunedin, Florida
  - Bayonet Point Hudson Kidney Center, Hudson, Florida
  - Outcomes Research International, Inc., Hudson, Florida
  - Bay Breeze Dialysis, Largo, Florida
  - New Port Richey Kidney Center, New Port Richey, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Nephrology consultants, Orlando, Florida
  - Hernando Kidney Center, Spring Hill, Florida
  - Nephrology Associates, P.C., Augusta, Georgia
  - MId Atlantic Nephrology Associates, PA, Baltimore, Maryland
  - Caritas St. Elizabeth Center, Boston, Massachusetts
  - Western New England Renal & Transplant Associatea, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Hypertension & Renal Research Group, Buffalo, New York
  - Bayview Nephrology, Inc., Erie, Pennsylvania
  - Kidney Associates, PLLC, Houston, Texas
  - Southwest Houston Research, LTD, Houston, Texas
  - Fox Valley Nephrology Associates, Appelton, Wisconsin

REFERENCES:
- [Derived] Maki DG, Ash SR, Winger RK, Lavin P; AZEPTIC Trial Investigators. A novel antimicrobial and antithrombotic lock solution for hemodialysis catheters: a multi-center, controlled, randomized trial. Crit Care Med. 2011 Apr;39(4):613-20. doi: 10.1097/CCM.0b013e318206b5a2. PMID 21200319